CLINICAL TRIAL: NCT05188040
Title: Virtual Reality in Hand Therapy Effectiveness and Implementation
Brief Title: Effectiveness of Virtual Reality in Hand Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Uhl (Other)
Collaborators: University of Kentucky (Other); Commonwealth Hand and Physical Therapy (Unknown)
Responsible Party: Sponsor-Investigator, Timothy Uhl, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72833
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Distal Radius Fracture; Chronic Regional Pain Syndrome; Flexor Tendon Rupture
Keywords: Virtual Reality; Function; Hand Therapy; Exercises
MeSH Terms: conditions — Wrist Fractures; Complex Regional Pain Syndromes; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Participants at the Commonwealth Hand and Physical Therapy clinic with the 3 included arm and hand injury diagnoses will be offered the opportunity in a flyer at the clinic to participate in the VR study. Those consented will complete the pre and post outcome measures outlined within this document with the research team member. For intervention, the participants will be instructed by the treating therapist in standard of care rehabilitation and utilize Virtual Reality with the Oculus Quest 2 system as the active exercise component of their rehabilitation over approximately approximately 4 sessions, totally ~ 1-hour. The specific virtual reality games within the Oculus Quest 2 VR system will be selected by the therapist providing interventions each session. The virtual reality game allows for augmented visual feedback and will be directly supervised by the treating therapists.
Masking Description: No Masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Intervention Group (Experimental): Hand Therapy Exercises utilizing Oculus Quest 2 VR system with augmented feedback for patient to perform active hand therapy. Specific interventions / games will be selected by the participants individual therapist.
  Interventions: Other: Virtual Reality Exercises

INTERVENTIONS:
Other: Virtual Reality Exercises — Hand Therapy Exercises utilizing Oculus Quest 2 VR system with augmented feedback for patient to perform active hand therapy. Specific interventions / games will be selected by the participants individual therapist.

SUMMARY:
The purpose of this study is to determine if the use of Virtual Reality as an intervention for patients following specific hand injuries will positively affect patients with decreased hand function and reduce pain and improve outcomes. Participants will be recruited from 3 different clinics in central Kentucky.

DETAILED DESCRIPTION:
Participants will participate in four sessions of therapy treatment over a 2-3 week time span of schedule therapy appointments during their active phase of rehabilitation for approximately 1-hour virtual reality (VR) training dosage which will be recorded. The specific virtual reality games within the Oculus Quest 2 VR system will be selected by the therapist providing interventions each session.

In addition to the Virtual Reality intervention noted above, participants will participate in a pre and post-test outcome measure session (25-30 minutes) with a research team member. (See outcome measure section for more details).

ELIGIBILITY:
Inclusion Criteria:

1. Attending hand therapy for rehabilitation of an upper extremity injury with a diagnosis of distal radius fracture, complex regional pain syndrome or tendon ruptures
2. Must be in an active exercise phase of rehabilitation

Exclusion Criteria:

1. Not in a phase in their rehabilitation in which they can perform active exercises
2. Having arm injury due to a neurological disorder (stroke, Multiple sclerosis, spinal cord injury, other)
3. Non-English speaking
4. Patient reporting a history of severe claustrophobia or motion sickness

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Hand Function Measures - Box and Block Test | 4 minutes
  The patient is asked to grasp a single block out of one box and move the block into the other box. They must cross midline to drop the box into the other box. This is a timed test for 1 minute. The number of blocks moved are counted and then the test is repeated with the other hand. A 15 second trial practice is performed so the participant understands the test. The number of blocks move with each hand is recorded.
Hand Function Measures - Nine Hole Peg Test | 8 minutes
  Nine Hole Peg Test measures finger dexterity and motor function. The participants will take 9 pegs from a container and place into a board as quickly as possible and then return them back to the container. A practice trial of this assessment will also occur prior to the documented time trial.

SECONDARY OUTCOMES:
Quick Disability of Arm Shoulder and Hand (QDASH) | 5 minutes
  Quick DASH (QDASH) subjective report measure is an 11-item questionnaire to indicate the level of disability a person is currently having given their injury. It is scored from 0-100 with 0 representing no disability and 100 indicating the have severe disability. A lower score is a better score on this outcome measure.
Visual Analog Scale | 1 minute
  Self-Report Pain Measure on a 0 - 10 scale.
Enjoyment Subscale of the Intrinsic Motivation Inventory scale | 7 minutes
  7 items on a subjective questionnaire (7 point Likert scale) - completed post intervention only

CONTACTS AND LOCATIONS:
Overall Officials: Tim L Uhl, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Commonwealth Hand and Physical Therapy, Georgetown, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tefertiller C, Hays K, Natale A, O'Dell D, Ketchum J, Sevigny M, Eagye CB, Philippus A, Harrison-Felix C. Results From a Randomized Controlled Trial to Address Balance Deficits After Traumatic Brain Injury. Arch Phys Med Rehabil. 2019 Aug;100(8):1409-1416. doi: 10.1016/j.apmr.2019.03.015. Epub 2019 Apr 19. PMID 31009598
- [Background] Palaus M, Marron EM, Viejo-Sobera R, Redolar-Ripoll D. Neural Basis of Video Gaming: A Systematic Review. Front Hum Neurosci. 2017 May 22;11:248. doi: 10.3389/fnhum.2017.00248. eCollection 2017. PMID 28588464
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Background] Cuthbert JP, Staniszewski K, Hays K, Gerber D, Natale A, O'Dell D. Virtual reality-based therapy for the treatment of balance deficits in patients receiving inpatient rehabilitation for traumatic brain injury. Brain Inj. 2014;28(2):181-8. doi: 10.3109/02699052.2013.860475. PMID 24456057
- [Background] Glegg SMN, Levac DE. Barriers, Facilitators and Interventions to Support Virtual Reality Implementation in Rehabilitation: A Scoping Review. PM R. 2018 Nov;10(11):1237-1251.e1. doi: 10.1016/j.pmrj.2018.07.004. PMID 30503231
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Fowler CA, Ballistrea LM, Mazzone KE, Martin AM, Kaplan H, Kip KE, Murphy JL, Winkler SL. A virtual reality intervention for fear of movement for Veterans with chronic pain: protocol for a feasibility study. Pilot Feasibility Stud. 2019 Dec 11;5:146. doi: 10.1186/s40814-019-0501-y. eCollection 2019. PMID 31890259
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Hoffman HG, Boe DA, Rombokas E, Khadra C, LeMay S, Meyer WJ, Patterson S, Ballesteros A, Pitt SW. Virtual reality hand therapy: A new tool for nonopioid analgesia for acute procedural pain, hand rehabilitation, and VR embodiment therapy for phantom limb pain. J Hand Ther. 2020 Apr-Jun;33(2):254-262. doi: 10.1016/j.jht.2020.04.001. Epub 2020 May 30. PMID 32482376